CLINICAL TRIAL: NCT06390189
Title: Inflammatory Resolution in Cardiometabolic Health and Disease - an Aarhus Based Cohort
Brief Title: Inflammatory Resolution in Cardiometabolic Health and Disease
Acronym: RESOLVE AU
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-102-23
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-04

CONDITIONS: Inflammation; Obesity; Cardiovascular Diseases
MeSH Terms: conditions — Inflammation; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Lean and metabolically healthy
- Lean and metabolically unhealthy
- Overweight and metabolically healthy
- Overweight and metabolically unhealthy
- Obese and metabolically healthy
- Obese and metabolically unhealthy

SUMMARY:
The specific aim of this study is to determine molecular pathways that differentiate metabolically healthy vs unhealthy human phenotypes, and to investigate the therapeutic potential of pro-resolving lipids. Investigators will recruit volunteers that are metabolically healthy or unhealthy that fall within three BMI ranges: lean (18.-24.9 kg/m2), overweight (25.0-29.9 kg/m2) and obese (>30.0 kg/m2). Investigators hypothesize that metabolically healthy individuals have a superior endogenous capacity to regulate an inflammatory/resolving response.

ELIGIBILITY:
Inclusion Criteria:

* Informed signed consent has been obtained from the volunteer.
* The volunteer has a BMI greater than 18.5 kg/m2
* Men and women over the age of 18 are included.

Exclusion Criteria:

* The study staff contacting a potential participant perceives that the individual has difficulty understanding the information.
* An MD determines that the individual is on too many medications to participate.
* The individual takes a medication that is approved by the MD, but he/she is not willing or not able to wait with any potential morning medication until after their fasted blood-draw.
* The individual states that they have increased bleeding tendency or are using anti-coagulant (blood thinning) medication.
* The individual has some form of chronic inflammation.
* The individual regularly uses medication that affects inflammatory resolution (e.g., low-dose aspirin).
* The individual uses immunosuppressive drugs (e.g., methotrexate).
* The individual regularly consumes fish oils (omega 3).
* The individual has significant gastrointestinal problems.
* The individual smokes or uses chewing tobacco.
* The individual has been drinking alcohol two days before the study visit.
* The individual has tattoos or body piercings on the forearms and / or the stomach that can affect the examination.
* The individual does not follow instructions given in the research study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals that contact the investigators (via phone or email) and express an interest in participating in the study will be invited to an information visit, after which the individual has at least 24 hours to consider their participation. For those that are interested in the study, the investigators then proceed to schedule visit 1-5.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Inflammation and resolution status measurements in different metabolic phenotypes | September 2028
  Quantifiable inflammatory resolution by measurement of IL-6 cytokine levels in the acute vs the resolving phase of blister formation.

SECONDARY OUTCOMES:
Systemic low-grade inflammation measurement in different phenotypes | September 2028
  Measurement of plasma C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No